CLINICAL TRIAL: NCT05615506
Title: Suction Diathermy Adenoidectomy : Efficacy and Safety
Brief Title: Suction Diathermy Adenoidectomy (SDA) : Efficacy and Safety
Acronym: SDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Hamed Hashem, principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-22-10-10
Record Dates: First submitted 2022-10-25; First posted 2022-11-14 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Adenoidectomy

STUDY DESIGN:
Intervention Model Description: patients under 15 years old who are scheduled to undergo elective adenoidectomy with or without ventilation tube application. , selected randomly, with symptoms and signs suggestive of adenoid hypertrophy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): suction diathermy adenoidectomy
  Interventions: Procedure: Suction Diathermy Adenoidectomy

INTERVENTIONS:
Procedure: Suction Diathermy Adenoidectomy — suction diathermy adenoidectomy

SUMMARY:
The aim of this prospective study is to evaluate the efficacy and safety of endoscopic suction diathermy adenoidectomy as regard the operative time, adenoid tissue remnant, blood loss, and clinical events like pain, halitosis, postoperative hemorrhage, speech changes and recurrence.

DETAILED DESCRIPTION:
Suction diathermy adenoidectomy is a procedure that uses thermal energy generated by electric current to ablate adenoid which is removed using suction. This procedure was described in 1997 and the technique has the advantage of complete tissue removal with reduced blood loss and intraoperative time, also reduced post-operative complications as postoperative hemorrhage , nasality and lower recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

1. Obstructive symptoms such as long-lasting nocturnal snoring, sleep apnea, and open mouth breathing, bilateral nasal obstruction, and/or bilateral nasal discharge.
2. Adenoid hypertrophy is the only cause of nasal obstruction.
3. Radiography evidence of adenoid hypertrophy encroaching on the airway column.
4. Age under 15 years.
5. Sex: both males and females.
6. All patients are generally well and fit for surgery.

Exclusion Criteria:

1. Presence of chronic diseases such as chronic heart diseases, chronic liver diseases, chronic renal diseases, and diabetes mellitus.
2. Patients with other causes of nasal obstruction such as acute rhinitis, allergic rhinitis, septal deviation, inferior turbinate hypertrophy, antrochoanal polyp, nasal polypi or anatomical deformities (Choanal atresia).
3. Cases with submucous cleft palate and cases with a previous history of cleft palate repair.
4. Patients with bleeding or coagulation defects.
5. Patients with atrophic rhinitis.
6. Patients with recurrent adenoid.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
the efficacy of suction diathermy in completeness of adenoid removal | intraoperative
  Flexible fibre optic nasopharyngoscope or zero degree nasal endoscope is used for evaluation of the nasopharynx and determine the adenoid remnant in percentage.
amount of intraoperative blood loss with suction diathermy adenoidectomy | intraoperative
  amount of blood loss measured in cubic centimeter
Recurrence of symptoms | 6 months
  Flexible fibre optic nasopharyngoscope or 0 degree nasal endoscope is used for evaluation of the nasopharynx to detect any remnant or recurrence of adenoid in percentage
postoperative hemorrhage | 2 weeks
  percentage of occurence of post operative hemorrhage

SECONDARY OUTCOMES:
Intraoperative trauma to adjacent structures with suction diathermy adenoidectomy | 6 months
  evaluated using zero degree nasal endoscope
Postoperative pain | 7 days
  pain is assessed using postoperative diary and pain is rated on a 0-10 visual analogue scale, 0 being no pain; and 10 being worse pain ever.
postoperative halitosis | 7 days
  halitosis is assessed using postoperative diary and halitosis is rated on 0-10 visual analogue scale, 0 being no odour, and 10 being the worst odour they have encountered
operative time with suction diathermy adenoidectomy | 6 months
  operative time measured in minutes
Speech changes | 6 months
  detection of open nasality and palatal assessment by Flexible fibre optic nasopharyngoscope after 3 weeks then 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Amr Hamed Hashem, Sohag, Egypt

REFERENCES:
- [Result] Gates GA, Muntz HR, Gaylis B. Adenoidectomy and otitis media. Ann Otol Rhinol Laryngol Suppl. 1992 Jan;155:24-32. doi: 10.1177/00034894921010s106. PMID 1728896
- [Result] Dinis PB, Haider H, Gomes A. The effects of adenoid hypertrophy and subsequent adenoidectomy on pediatric nasal airway resistance. Am J Rhinol. 1999 Sep-Oct;13(5):363-9. doi: 10.2500/105065899781367564. PMID 10582114
- [Result] Clemens J, McMurray JS, Willging JP. Electrocautery versus curette adenoidectomy: comparison of postoperative results. Int J Pediatr Otorhinolaryngol. 1998 Mar 1;43(2):115-22. doi: 10.1016/s0165-5876(97)00159-6. PMID 9578120
- [Result] Shapiro NL, Bhattacharyya N. Cold dissection versus coblation-assisted adenotonsillectomy in children. Laryngoscope. 2007 Mar;117(3):406-10. doi: 10.1097/MLG.0b013e31802ffe47. PMID 17334301
- [Result] Pagella F, Pusateri A, Canzi P, Caputo M, Marseglia A, Pelizzo G, Matti E. The evolution of the adenoidectomy: analysis of different power-assisted techniques. Int J Immunopathol Pharmacol. 2011 Oct;24(4 Suppl):55-9. doi: 10.1177/03946320110240S411. PMID 22032788
- [Result] Wright ED, Manoukian JJ, Shapiro RS. Ablative adenoidectomy: a new technique using simultaneous liquefaction/aspiration. J Otolaryngol. 1997 Feb;26(1):36-43. PMID 9055172
- [Result] Regmi D, Mathur NN, Bhattarai M. Rigid endoscopic evaluation of conventional curettage adenoidectomy. J Laryngol Otol. 2011 Jan;125(1):53-8. doi: 10.1017/S0022215110002100. Epub 2010 Oct 18. PMID 20950511
- [Result] Agrawal V, Agarwal PK, Agrawal A. Defining the Surgical Limits of Adenoidectomy so as to Prevent Recurrence of Adenoids. Indian J Otolaryngol Head Neck Surg. 2016 Jun;68(2):131-4. doi: 10.1007/s12070-016-0971-7. Epub 2016 Mar 12. PMID 27340625